CLINICAL TRIAL: NCT07223528
Title: A Phase 2a Single Arm Open Label Safety and Efficacy Study of Telaglenastat Plus Standard of Care in Adults With Functional Class Ii-iii Precapillary Pulmonary Hypertension Across Wsph Groups 1-4
Brief Title: TEPH: Telaglenastat Efficacy in Pulmonary Hypertension
Acronym: TEPH
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chan, Stephen, MD, PhD (Other)
Collaborators: Synhale Theraputics (Unknown)
Responsible Party: Principal Investigator, Michael Risbano, Assistant Professor of Medicine, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY24070041
Record Dates: First submitted 2025-10-21; First posted 2025-11-03 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Hypertension
Keywords: pulmonary hypertension; lung disease; telaglenastat
MeSH Terms: conditions — Hypertension, Pulmonary; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Open-Label Telaglenastat Arm (Experimental)
  Interventions: Drug: Telaglenastat

INTERVENTIONS:
Drug: Telaglenastat — The participant will need to come in for a screening visit prior prescribing the medication to confirm eligibility. The visit will include physical exams, labs, right heart cath, and maybe pulmonary function test and chest imaging. Eligible participants will be taking 800 mg Telaglenastat (CB-839) by mouth with food twice a day for a total of 12 weeks. Participants will need to come in for study related visits during this time. At the end of 12 months period, we will need to repeat same activities we did prior to prescribing to medication. Pending FDA approval, eligible participants may continue Telaglenastat for an additional 12 weeks.

SUMMARY:
The research study is being conducted to evaluate the effectiveness of a drug called Telaglenastat in adults diagnosed with Pulmonary Hypertension (PH). PH is a progressive condition that affects the arteries in the lungs, specifically the pulmonary arteries, which carry blood from the right side of the heart to the lungs. Telaglenastat is not currently approved by the Food and Drug Administration for the treatment of PH. However, the study investigators believe that Telaglenastat may help lower blood pressure in the lungs and improve both heart and lung function. It is important to note that the drug will not be available to participants once the study concludes.

DETAILED DESCRIPTION:
The study will consist of the following visits:

1. Screening Visit (30-60 mins)

   * Consenting
   * Medical history, physical exam, lab tests (blood, urine)
   * Review of past heart/lung records
   * Surveys
2. Baseline Visit (Visit 2, 2-3 hrs)

   * Physical exam, 6-minute walk test
   * Echo, Right Heart Catheterization (RHC)
   * High-Resolution CT (HRCT) & Pulmonary Function Tests (PFTs) if applicable
   * Lab tests, ECG, glutamine blood sample
   * Surveys
3. Treatment Phase (Visits 3-6, Weeks 1,2,4,8) Telaglenastat 800 mg/twice daily

   Short visits (30 mins) for:
   * Physical Exam
   * Surveys
   * Labs
4. Visit 7 End of Treatment (week 12, 2-3 hours) include the following:

   * Physical Exam
   * 6 Minute Walk Test
   * Echo/RHC/ECG
   * HRCT/PFT group 3
   * Labs
   * Surveys

     * Optional Extension (Visits 8-12, Weeks 13-24) Same procedures as initial 12 weeks Final visit includes full reassessment

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18-75 years old.
2. Able to provide written informed consent.
3. Able to comply with study procedures, able to undergo cardiac catheterization and exercise testing.
4. Patients will be identified with PH Group 1-4 PH by an expert clinician in the UPMC Comprehensive Care Center for Pulmonary Hypertension.
5. For Group 1, 3, and 4 PH, prior right heart catheterization (RHC) should show documented diagnosis of precapillary PH at mean pulmonary arterial pressure (mPAP > 20 mm Hg, PCWP < 15 mm Hg, and PVR > 4 WU) within 1 year of randomization. If patient doesn't have RHC within 1 year, we will repeat RHC at baseline visit. For Group 2 PH, prior right heart catheterization (RHC) should show mean pulmonary arterial pressure mPAP > 20 mm Hg and PVR > 4 WU within one year of randomization. If patient don't have RHC within 1 year we will repeat RHC at baseline visit.
6. Minimum pulmonary vascular resistance (PVR) of > 4 Wood units by RHC at screening within last 6 months on at least one month of stable medical therapy.
7. Symptomatic PH classified as WHO functional class II or III.
8. Body mass index (BMI) 18 to 40 kg/m² at Screening. If BMI is > 35 kg/m², subject chest circumference should be < 65 inches (165 cm).
9. 6-minute walk distance (6MWD) ≥ 100 meters (m) and < 550 m at screening.
10. For Group 1 PH, patients on SOC medical treatment for PH with vasodilators or Sotatercept are required to have been receiving a stable dose for at least 3 months before undergoing randomization.
11. For Group 2 PH-HFpEF: Documented transthoracic echocardiogram or cardiac MRI with LV ejection fraction > 50% within 6 months of enrollment, along with meeting at least one of the three criteria by echocardiographic/MRI: (1) Diastolic dysfunction, (2) Left atrial enlargement (LA diameter > 3.6 cm), or (3) Prior right heart catheterization data indicating PCWP > 15 mm Hg. Stable heart failure therapy for at least 30 days.
12. For Group 3 PH-ILD, documented diagnosis of interstitial lung disease (diffuse parenchymal lung disease) by high resolution lung CT scan within 6 months of randomization. Patients with Group 3 PH with connective tissue disease should have confirmed baseline FVC < 70% within 6 months of randomization. For subjects with a history of lobectomy or pneumonectomy, and for whom there are no population-based normalization methods, assessment based on residual lung volume will be permitted to assess eligibility. Patients receiving drug treatment (i.e., pirfenidone or nintedanib) for their underlying lung disease or pulmonary hypertension (i.e., inhaled Treprostinil) should receive a stable dose for at least 30 days before undergoing randomization.
13. For Group 4 PH (CTEPH) eligible patients will have V/Q scan or CT scan with contrast demonstrating chronic thromboembolic disease in the pulmonary vasculature at least 6 months after most recent pulmonary embolus and with right heart catheterization within one year of enrollment. If patient doesn't have RHC within 1 year, we will repeat RHC at baseline visit. Eligible patients will include those with inoperable CTEPH or at least 6 months post-surgery with persistent thromboembolic disease. Patients receiving approved therapies for pulmonary hypertension are required to have been receiving a stable dose for at least 30 days before undergoing randomization.
14. Women of childbearing potential must be willing and able to practice medically acceptable effective contraception during the study and continuing contraception for 30 days after their last dose of study drug. Women who are surgically sterile or those who are post-menopausal for at least 2 years are not considered to be of childbearing potential. Men who are not sterile must also agree to use contraception.

Exclusion Criteria:

1. For Group 2 PH-HFpEF patients:

   * With clinically decompensated heart failure
   * Uncontrolled hypertension (SBP > 160 mm Hg, DBP > 90)
   * Echocardiographic/MRI
   * Evidence of moderate-severe mitral regurgitation or mitral stenosis within 6 months of enrollment
2. Group 3 PH-ILD, patients receiving approved therapies other than inhaled Treprostinil for PAH within 60 days before randomization are not eligible for enrollment.
3. Group 1 PH, patients naïve to medical treatment for PH are not eligible for enrollment.
4. History of lung reduction surgery or likely to undergo lung transplantation within the next 6 months.
5. Enrolled in, or planned participation in, device or other interventional clinical studies or cardio-pulmonary rehabilitation programs, based upon exercise within 90 days of Screening or during study participation.
6. Patients with other secondary causes of PH including, but not limited to, left or right heart failure, valvular heart disease, chronic obstructive lung disease, atrial septal defect with left to right shunt, and sleep apnea will be excluded if it was the primary cause of PAH.
7. Diagnosed with significant (≥ 2+ regurgitation) mitral regurgitation or aortic regurgitation valvular disease
8. Uncontrolled hypertension (SBP > 160 mm Hg, DBP > 90)
9. Left ventricular ejection fraction (LVEF) < 45%
10. Adult congenital heart disease (ACHD)
11. Sustained systolic blood pressure (SBP) < 95 mmHg and/or diastolic blood pressure (DBP) < 50 mmHg (confirmed by duplicate seated readings) on at least 3 consecutive occasions (self-monitored or office) prior to or at Screening, or overt symptomatic hypotension
12. Sustained resting heart rate (HR) > 120 beats per minute (confirmed by duplicate assessments of office vital signs) or consecutive electrocardiogram (ECG) assessments on at least 3 consecutive occasions prior to or at Screening
13. Concomitant medical or psychiatric disorder, condition, history, or any other condition that, in the opinion of the Investigator, would either put the participant at risk or impair their ability to participate in or complete the requirements of the study or confound the objectives of the study
14. Concomitant medical disorder that is expected to limit the subject's life-expectancy to ≤ 1 year
15. Untreated, moderate to severe obstructive sleep apnea
16. Evidence of thrombocytopenia (platelets < 150,000/mm³), significant chronic thromboembolic disorder, or recent pulmonary embolism within 6 months prior to Screening
17. History of a bleeding disorder
18. Known porphyria, mitochondrial, or urea cycle disease
19. History of chronic pancreatic disease
20. Pregnant or lactating female
21. Active coronavirus disease 19 (COVID-19); however, those with previous COVID-19 are permitted
22. Participated in another investigational drug study within 30 days prior to Screening or is participating in a non-medication study which, in the opinion of the Investigator, would interfere with the study compliance or outcome assessments
23. Glomerular Filtration Rate (GFR) of < 30 mL/min/1.73m²
24. Significant liver dysfunction as measured by any one of the following at Screening (including subjects with acute or chronic hepatitis as well as subjects with own or family history of serious hepatitis, especially drug related):

    * Alanine aminotransferase (ALT) > 2.0 × upper limit of normal (ULN)
    * Aspartate aminotransferase (AST) > 2.0 × ULN
    * Serum bilirubin ≥ 1.6 mg/dL or > 2.0 × ULN
25. Known history of substance abuse including alcohol abuse within the 1 year prior to Screening that in the opinion of the Investigator would impair the subject's ability to participate in or complete the requirements of the study
26. Any major surgical procedure or trauma within 30 days prior to Screening or planned surgical procedure during the study period.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-09-25 (Estimated); Study Completion 2028-09-25 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular Resistance (PVR) measured via Right Hearth Catheterization (RHC) | Visit 2 at week 1 and Visit 7 at week 12
  We will use PVR to measure the effect of treatment on PH

SECONDARY OUTCOMES:
Functional class (FC) | The functional class will be determined at week 1 and 12
  We will use the functional class evaluated by licensed physician based on clinical history.
  Functional Class I: No symptoms with normal activity. Class II: Mild symptoms with ordinary activity (e.g., walking, climbing stairs).
  Class III: Noticeable symptoms with less-than-ordinary activity; limited daily tasks.
  Class IV: Symptoms at rest; unable to perform any physical activity without discomfort.
6 minute walk test | 6MWT will be at week 1 and 12
  The person walks back and forth along a marked corridor for 6 minutes. They can slow down, stop, or rest if needed. The total distance walked is recorded in meters. Will be completed by clinical research coordinator
NT-proBNP | Will be measure at week 1 and 12
  Blood work including NT-proBNP will be drawn by CRC
Glutamine and glutamate plasma levels | Will be done on screening visit, on week 1 and week 12
  Measure serum glutamine/glutamate ratio

CONTACTS AND LOCATIONS:
Overall Officials: Michael Risbano, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presybeterian, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with other individuals for future research and if shared will be shared without identifiers.
  Participant's medical record information contained within the Research study may be provided to secondary research investigators (i.e., research investigators who are not affiliated with the Comprehensive Pulmonary Hypertension Program at University of Pittsburgh).The type of data shared would include demographic information, past medical history, medications, lab results, right heart Cath hemodynamics and cardiac imaging studies. However, prior to its provision to any secondary investigators, the information shall be de-identified. The Comprehensive Pulmonary Hypertension Program and Comprehensive lung center shall require secondary investigators to obtain regulatory approval prior its provision of de-identified information to the secondary investigators.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will available starting 6 months after publication
Access Criteria: The Comprehensive Pulmonary Hypertension Program and Comprehensive lung center shall require secondary investigators to obtain regulatory approval prior its provision of de-identified information to the secondary investigators